CLINICAL TRIAL: NCT00831662
Title: The Effects of Diquafosol Tetrasodium Ophthalmic Solution, 2% in Subjects With Dry Eye Disease (P08637)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P08637; 03-113
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2014-12

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 1 (Experimental)
  Interventions: Drug: Diquafosol tetrasodium ophthalmic solution, 2%

INTERVENTIONS:
Drug: Diquafosol tetrasodium ophthalmic solution, 2% — One to two drops in each eye QID for 6 weeks
  Arms: Arm 1
Drug: Placebo — One to two drops in each eye QID for 6 weeks
  Arms: Arm 2

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of diquafosol tetrasodium ophthalmic solution, 2% vs. placebo, in subjects with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Have best corrected visual acuity in both eyes of at least +0.7 or better
* Central corneal staining of 3 on the NEI scale
* If female, are non-pregnant or non-lactating
* Have a history of dry eye disease in both eyes
* Have normal lid anatomy

Exclusion Criteria:

* Unable to withhold the use of contact lenses during the study or 2 weeks prior to the study
* Have had ocular surface surgery within the past year
* Are considered legally blind in one eye
* Have a serious medical condition which could confound study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects that achieve clearing of fluorescein staining of the central cornea (NEI scale). Subjects must have a score of 0 on the NEI scale at Week 6 to be considered responders. | 6 weeks

SECONDARY OUTCOMES:
Proportion of subjects that achieve a 2-or-more-unit reduction of fluorescein staining of the central cornea (NEI scale) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD, PhD, Study Director — Medical Monitor, Inspire

REFERENCES:
- [Result] Tauber J, Davitt WF, Bokosky JE, Nichols KK, Yerxa BR, Schaberg AE, LaVange LM, Mills-Wilson MC, Kellerman DJ. Double-masked, placebo-controlled safety and efficacy trial of diquafosol tetrasodium (INS365) ophthalmic solution for the treatment of dry eye. Cornea. 2004 Nov;23(8):784-92. doi: 10.1097/01.ico.0000133993.14768.a9. PMID 15502479